CLINICAL TRIAL: NCT00277745
Title: Integrated Microfluidic System for Oral Diagnostics
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Sandia National Laboratories (Industry); National Institutes of Health (NIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, William Giannobile, William Giannobile, D.D.S., D.Med.Sc., University of Michigan
Other Study IDs: H03-00003522; U01DE014961-01 (NIH)
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Healthy; Periodontitis
Keywords: periodontitis; microfluidics; saliva diagnostics
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva, serum, dental plaque and gingival crevicular fluid
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: miniaturized microfluidic system — Subjects will provide appropriate periodontal treatment as needed.

SUMMARY:
This study is being conducted to test the ability and accuracy of a new instrument in the diagnosis of periodontitis (gum disease) by using fluids from the mouth. The diagnosis instrument will test two types of fluids, gingival crevicular fluid (GCF) and saliva. GCF is the fluid that accumulates between your teeth and gum tissue. The fluids will be collected in three ways: 1. Direct GCF sampling 2. GCF rinse sampling and 3. Whole saliva. A total of 100 adult patients will participate in this study. These subjects will be of two patient populations: 1) diseased population, with active gum disease; and 2) a low-risk disease population, with no active gum disease. Patients will be seen 6 times over the course of the study over a period of approximately 12 months. At each visit the patient will undergo oral fluid collection, as previously described, and thorough examinations of the mouth, including the taking of measurements for study purposes. Patients will also have radiographs taken at baseline, month 6, and end of study visits.

DETAILED DESCRIPTION:
The ultimate goal of this investigation is to validate the ability of the prototype platform (miniaturized microfluidic device that can rapidly (within 15 minutes) measure small volumes of oral fluids (on the order of nanoliters of fluid) and identify biomarkers of disease such as mediators of inflammation (interleukins -1 and -6; C-reactive protein (CRP), and a marker of bone resorption (ICTP). This analysis will aid in the diagnosis of active periodontal (gum) disease as well as diseases involved in systemic inflammation (e.g., cardiovascular disease) or systemic bone loss (osteoporosis). This project will have two specific goals: 1. To validate the ability of the diagnostic to measure the designated mediators from oral fluids; and 2. Determine the ability of the multiplexed format of mediator analysis to predict disease activity (future bone loss) in patients at high and low risk for disease. This proposed feasibility study will then aid in providing the impetus for sample size and other design requirements for larger, more expanded human clinical trial testing and subsequent technology transfer.

ELIGIBILITY:
Inclusion Criteria:

* Must possess at least 20 teeth and not have received periodontal treatment or antibiotic-related therapy for medical or dental reasons 3 months prior to study inclusion.
* Low-risk inclusion: < 3 mm of attachment loss, no pockets > 4 mm, possess no radiographic bone loss, and < 20 sites with bleeding on probing (BOP). Low-risk cohort will be comprised of at least > 50% of the subjects above age 35 in order to exam low risk patients in other age strata (so as to decrease potential bias towards a younger population in the low risk cohort).
* Disease-susceptible inclusion: Exhibit at least 4 sites with evidence of radiographic bone loss, mean attachment loss > 3 mm, pocket depths (PD) > 4 mm and BOP.

Exclusion Criteria:

* Long-term use of medications known to affect periodontal status such as anti-inflammatory drugs (NSAIDS and aspirins)
* History of metabolic bone diseases such as rheumatoid arthritis or post-menopausal osteoporosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 Adult subjects comprised of two populations: 1) disease susceptible (n=50) and 2) low-risk disease (n=50)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2005-06; Primary Completion 2007-02 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Proof of principle study to determine ability of device to predict disease activity in patients at high and low risk for disease. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: William V Giannobile, DDS, DMedSc, Principal Investigator — Director of MCOHR
Locations (1):
- Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Herr AE, Hatch AV, Giannobile WV, Throckmorton DJ, Tran HM, Brennan JS, Singh AK. Integrated microfluidic platform for oral diagnostics. Ann N Y Acad Sci. 2007 Mar;1098:362-74. doi: 10.1196/annals.1384.004. PMID 17435142
- [Background] Kinney JS, Ramseier CA, Giannobile WV. Oral fluid-based biomarkers of alveolar bone loss in periodontitis. Ann N Y Acad Sci. 2007 Mar;1098:230-51. doi: 10.1196/annals.1384.028. PMID 17435132
- [Result] Ramseier CA, Kinney JS, Herr AE, Braun T, Sugai JV, Shelburne CA, Rayburn LA, Tran HM, Singh AK, Giannobile WV. Identification of pathogen and host-response markers correlated with periodontal disease. J Periodontol. 2009 Mar;80(3):436-46. doi: 10.1902/jop.2009.080480. PMID 19254128
- [Result] Sweier DG, Shelburne PS, Giannobile WV, Kinney JS, Lopatin DE, Shelburne CE. Immunoglobulin G (IgG) class, but Not IgA or IgM, antibodies to peptides of the Porphyromonas gingivalis chaperone HtpG predict health in subjects with periodontitis by a fluorescence enzyme-linked immunosorbent assay. Clin Vaccine Immunol. 2009 Dec;16(12):1766-73. doi: 10.1128/CVI.00272-09. Epub 2009 Sep 30. PMID 19793900
- [Result] Kinney JS, Morelli T, Braun T, Ramseier CA, Herr AE, Sugai JV, Shelburne CE, Rayburn LA, Singh AK, Giannobile WV. Saliva/pathogen biomarker signatures and periodontal disease progression. J Dent Res. 2011 Jun;90(6):752-8. doi: 10.1177/0022034511399908. Epub 2011 Mar 15. PMID 21406610
- [Result] Kinney JS, Morelli T, Oh M, Braun TM, Ramseier CA, Sugai JV, Giannobile WV. Crevicular fluid biomarkers and periodontal disease progression. J Clin Periodontol. 2014 Feb;41(2):113-120. doi: 10.1111/jcpe.12194. Epub 2013 Dec 12. PMID 24303954